CLINICAL TRIAL: NCT01067521
Title: A Multinational, Multicenter, Randomized, Parallel-group Study Performed in Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS) to Assess the Efficacy, Safety and Tolerability of Glatiramer Acetate (GA) Injection 40 mg Administered Three Times a Week Compared to Placebo in a Double-blind Design
Brief Title: A Study in Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS) to Assess the Efficacy, Safety and Tolerability of Glatiramer Acetate (GA) Injection 40 mg Administered Three Times a Week Compared to Placebo
Acronym: GALA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-GA-301; 2009-018084-27 (EudraCT Number)
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; Glatiramer Acetate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GA 40 mg / GA 40 mg (Experimental): Also referred to as the 'Early Start' treatment arm, participants were administered glatiramer acetate (GA) 40 mg/mL by subcutaneous injection three times a week for 12 months during the Double-Blind Period, and then continued that treatment as open-label therapy until the drug was commercially available or development stopped.
  Interventions: Drug: Glatiramer acetate (GA)
- Placebo / GA 40 mg (Placebo Comparator): Also referred to as the 'Delayed Start' treatment arm, participants were administered placebo subcutaneous injections three times a week for 12 months during the Double-Blind Period, and then switched to GA 40 mg/mL subcutaneous injections three times a week as open-label therapy until the drug was commercially available or development stopped.
  Interventions: Drug: Glatiramer acetate (GA); Drug: Placebo

INTERVENTIONS:
Drug: Glatiramer acetate (GA) — GA 40 mg/mL administered 3 times a week by subcutaneous injection for a period of 12 months for participants assigned to GA treatment in the Double-Blind Period, and GA 40 mg/mL administered 3 times a week by subcutaneous injection for all participants in the Open-Label Extension Period.
  Other Names: Copaxone
Drug: Placebo — Placebo comparator administered by subcutaneous injection three times each week for 12 months during the Double-Blind Period.
  Arms: Placebo / GA 40 mg

SUMMARY:
The study is designed to assess the efficacy of Glatiramer Acetate (GA) injection 40 mg administered three times a week compared to placebo in subjects with RRMS, as measured by the number of confirmed relapses during the 12 month placebo controlled period. The study has two periods:

* Placebo Controlled Period: 12 months of 40 mg administered three times a week by subcutaneous injection or matching placebo.
* Open Label Extension Period: All subjects will continue treatment with GA 40 mg administered three times a week, until this dose strength is commercially available for the treatment of relapsing remitting multiple sclerosis (RRMS) patients or until the development of this GA dose regimen is stopped by the Sponsor

DETAILED DESCRIPTION:
Participants who were randomized to the GA 40 mg treatment arm in the Double-Blind Period, continue that treatment in the Open-Label Extension Period and are referred to as "Early Start" participants. Participants randomized to the Placebo arm in the Double-Blind Period and switched to GA 40 mg subcutaneous injections three times a week in the Open-Label Extension are referred to as "Delayed Start" participants.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a confirmed and documented MS diagnosis as defined by the Revised McDonald criteria with a relapsing-remitting disease course.
2. Subjects must be ambulatory with an EDSS score of 0-5.5 in both screening and baseline visits.
3. Subjects must be in a relapse-free, stable neurological condition and free of corticosteroid treatment [intravenous (IV), intramuscular (IM) and/or per os (PO)] or ACTH 30 days prior to screening (month -1) and between screening and baseline (month 0) visits.
4. Subjects must have experienced one of the following:

   At least one documented relapse in the 12 months prior to screening, or At least two documented relapses in the 24 months prior to screening, or One documented relapse between 12 and 24 months prior to screening with at least one documented T1-Gd enhancing lesion in an MRI performed within 12 months prior to screening.
5. Subjects must be between 18 and 55 years of age, inclusive.
6. Women of child-bearing potential must practice an acceptable method of birth control.
7. Subjects must be able to sign and date a written informed consent prior to entering the study.
8. Subjects must be willing and able to comply with the protocol requirements for the duration of the study

Exclusion Criteria:

1. Subjects with progressive forms of MS.
2. Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to screening.
3. Use of immunosuppressive (including Mitoxantrone and Fingolimod) or cytotoxic agents within 6 months prior to the screening visit.
4. Use of natalizumab (Tysabri®) or any other monoclonal antibodies within 2 years prior to screening.
5. Use of cladribine within 2 years prior to screening.
6. Previous treatment with immunomodulators (including IFNβ 1a and 1b, and IV Immunoglobulin (IVIg) within 2 months prior to screening.
7. Previous use of GA or any other glatiramoid.
8. Chronic (more than 30 consecutive days) systemic (IV, PO or IM) corticosteroid treatment within 6 months prior to screening visit.
9. Previous total body irradiation or total lymphoid irradiation.
10. Previous stem-cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
11. Pregnancy or breastfeeding.
12. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical exams, ECG, abnormal laboratory tests and chest X-ray. Such conditions may include hepatic, renal or metabolic diseases, systemic disease, acute infection, current malignancy or recent history (5 years) of malignancy, major psychiatric disorder, history of drug and/or alcohol abuse and allergies that could be detrimental according to the investigator's judgment.
13. A known history of sensitivity to Gadolinium.
14. Inability to successfully undergo MRI scanning.
15. A known drug hypersensitivity to Mannitol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1404 (Actual)
Dates: Start 2010-06-22 (Actual); Primary Completion 2012-05-08 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (176):
- United States (37):
  - Teva Investigational Site 1332, Birmingham, Alabama
  - Teva Investigational Site 1327, Gilbert, Arizona
  - Teva Investigational Site 1311, Phoenix, Arizona
  - Teva Investigational Site 1326, Fullerton, California
  - Teva Investigational Site 1335, La Jolla, California
  - Teva Investigational Site 1297, Aurora, Colorado
  - Teva Investigational Site 1344, Boulder, Colorado
  - Teva Investigational Site 1315, Centennial, Colorado
  - Teva Investigational Site 1350, Fort Collins, Colorado
  - Teva Investigational Site 1345, Miami, Florida
  - Teva Investigational Site 1336, Naples, Florida
  - Teva Investigational Site 1347, Pompano Beach, Florida
  - Teva Investigational Site 1319, Ponte Vedra, Florida
  - Teva Investigational Site 1298, Sarasota, Florida
  - Teva Investigational Site 1316, Sarasota, Florida
  - Teva Investigational Site 1340, Tampa, Florida
  - Teva Investigational Site 1317, Vero Beach, Florida
  - Teva Investigational Site 1303, Northbrook, Illinois
  - Teva Investigational Site 1334, Lenexa, Kansas
  - Teva Investigational Site 1302, Lexington, Kentucky
  - Teva Investigational Site 1322, Shreveport, Louisiana
  - Teva Investigational Site 1306, Detroit, Michigan
  - Teva Investigational Site 1329, Akron, Ohio
  - Teva Investigational Site 1349, Columbus, Ohio
  - Teva Investigational Site 1313, Dayton, Ohio
  - Teva Investigational Site 1318, Uniontown, Ohio
  - Teva Investigational Site 1341, Oklahoma City, Oklahoma
  - Teva Investigational Site 1310, Nashville, Tennessee
  - Teva Investigational Site 1321, Lubbock, Texas
  - Teva Investigational Site 1337, Round Rock, Texas
  - Teva Investigational Site 1301, San Antonio, Texas
  - Teva Investigational Site 1346, San Antonio, Texas
  - Teva Investigational Site 1343, Salt Lake City, Utah
  - Teva Investigational Site 1338, Richmond, Virginia
  - Teva Investigational Site 1339, Roanoke, Virginia
  - Teva Investigational Site 1300, Vienna, Virginia
  - Teva Investigational Site 1323, Kirkland, Washington
- Bulgaria (20):
  - Teva Investigational Site 5940, Blagoevgrad
  - Teva Investigational Site 5931, Pleven
  - Teva Investigational Site 5932, Pleven
  - Teva Investigational Site 5933, Plovdiv
  - Teva Investigational Site 5936, Rousse
  - Teva Investigational Site 5935, Shumen
  - Teva Investigational Site 5939, Sofia
  - Teva Investigational Site 5921, Sofia
  - Teva Investigational Site 5922, Sofia
  - Teva Investigational Site 5926, Sofia
  - Teva Investigational Site 5938, Sofia
  - Teva Investigational Site 5924, Sofia
  - Teva Investigational Site 5927, Sofia
  - Teva Investigational Site 5923, Sofia
  - Teva Investigational Site 5925, Sofia
  - Teva Investigational Site 5928, Sofia
  - Teva Investigational Site 5929, Sofia
  - Teva Investigational Site 5934, Stara Zagora
  - Teva Investigational Site 5930, Varna
  - Teva Investigational Site 5937, Veliko Tarnovo
- Croatia (5):
  - Teva Investigational Site 6011, Osijek
  - Teva Investigational Site 6009, Zagreb
  - Teva Investigational Site 6010, Zagreb
  - Teva Investigational Site 6012, Zagreb
  - Teva Investigational Site 6013, Zagreb
- Czechia (4):
  - Teva Investigational Site 5433, Olomouc
  - Teva Investigational Site 5434, Ostrava - Poruba
  - Teva Investigational Site 5432, Prague
  - Teva Investigational Site 5435, Teplice
- Estonia (3):
  - Teva Investigational Site 5513, Kohtla-Järve
  - Teva Investigational Site 5510, Tallinn
  - Teva Investigational Site 5512, Tartu
- Georgia (2):
  - Teva Investigational Site 8110, Tbilisi
  - Teva Investigational Site 8111, Tbilisi
- Germany (15):
  - Teva Investigational Site 3268, Bad Wildbad
  - Teva Investigational Site 3272, Bayreuth
  - Teva Investigational Site 3262, Berlin
  - Teva Investigational Site 3276, Berlin
  - Teva Investigational Site 3271, Bonn
  - Teva Investigational Site 3265, Dresden
  - Teva Investigational Site 3267, Düsseldorf
  - Teva Investigational Site 3263, Erbach im Odenwald
  - Teva Investigational Site 3269, Hamburg
  - Teva Investigational Site 3266, Hanover
  - Teva Investigational Site 3270, Herborn
  - Teva Investigational Site 3273, Kaltenkirchen
  - Teva Investigational Site 3275, Marburg
  - Teva Investigational Site 3261, Münster
  - Teva Investigational Site 3264, Ulm
- Hungary (7):
  - Teva Investigational Site 5127, Budapest
  - Teva Investigational Site 5129, Debrecen
  - Teva Investigational Site 5130, Eger
  - Teva Investigational Site 5132, Esztergom
  - Teva Investigational Site 5131, Győr
  - Teva Investigational Site 5128, Kaposvár
  - Teva Investigational Site 5133, Veszprém
- Teva Investigational Site 8052, Ramat Gan, Israel
- Italy (5):
  - Teva Investigational Site 3089, Bologna
  - Teva Investigational Site 3084, Cefalù
  - Teva Investigational Site 3092, Cosenza
  - Teva Investigational Site 3080, Milan
  - Teva Investigational Site 3086, Rome
- Lithuania (3):
  - Teva Investigational Site 5710, Kaunas
  - Teva Investigational Site 5712, Šiauliai
  - Teva Investigational Site 5711, Vilnius
- Poland (18):
  - Teva Investigational Site 5374, Częstochowa
  - Teva Investigational Site 5377, Elblag
  - Teva Investigational Site 5381, Gdansk
  - Teva Investigational Site 5380, Gdansk
  - Teva Investigational Site 5382, Gmina Końskie
  - Teva Investigational Site 5376, Gorzów Wielkopolski
  - Teva Investigational Site 5372, Grodzisk Mazowiecki
  - Teva Investigational Site 5375, Katowice
  - Teva Investigational Site 5368, Katowice
  - Teva Investigational Site 5379, Kielce
  - Teva Investigational Site 5369, Kościerzyna
  - Teva Investigational Site 5378, Krakow
  - Teva Investigational Site 5366, Lodz
  - Teva Investigational Site 5373, Olsztyn
  - Teva Investigational Site 5384, Poznan
  - Teva Investigational Site 5371, Szczecin
  - Teva Investigational Site 5367, Warsaw
  - Teva Investigational Site 5370, Wroclaw
- Romania (14):
  - Teva Investigational Site 5233, Baloteşti
  - Teva Investigational Site 5222, Bucharest
  - Teva Investigational Site 5221, Bucharest
  - Teva Investigational Site 5220, Bucharest
  - Teva Investigational Site 5227, Cluj-Napoca
  - Teva Investigational Site 5230, Cluj-Napoca
  - Teva Investigational Site 5225, Constanța
  - Teva Investigational Site 5226, Constanța
  - Teva Investigational Site 5232, Craiova
  - Teva Investigational Site 5231, Iași
  - Teva Investigational Site 5223, Piatra Neamţ
  - Teva Investigational Site 5228, Sibiu
  - Teva Investigational Site 5229, Târgu Mureş
  - Teva Investigational Site 5224, Timișoara
- Russia (17):
  - Teva Investigational Site 5063, Barnaul
  - Teva Investigational Site 5068, Irkutsk
  - Teva Investigational Site 5067, Krasnoyarsk
  - Teva Investigational Site 5052, Moscow
  - Teva Investigational Site 5057, Nizhny Novgorod
  - Teva Investigational Site 5062, Novosibirsk
  - Teva Investigational Site 5060, Perm
  - Teva Investigational Site 5056, Saint Petersburg
  - Teva Investigational Site 5055, Saint Petersburg
  - Teva Investigational Site 5053, Saint Petersburg
  - Teva Investigational Site 5054, Saint Petersburg
  - Teva Investigational Site 5058, Samara
  - Teva Investigational Site 5064, Smolensk
  - Teva Investigational Site 5066, Tomsk
  - Teva Investigational Site 5061, Ufa
  - Teva Investigational Site 5065, Yaroslavl
  - Teva Investigational Site 5059, Yekaterinburg
- South Africa (7):
  - Teva Investigational Site 9020, Johannesburg
  - Teva Investigational Site 9019, Johannesburg
  - Teva Investigational Site 9022, Pietermaritzburg
  - Teva Investigational Site 9025, Pretoria
  - Teva Investigational Site 9018, Pretoria
  - Teva Investigational Site 9021, Rosebank
  - Teva Investigational Site 9024, Umhlanga
- Ukraine (15):
  - Teva Investigational Site 5835, Chernihiv
  - Teva Investigational Site 5834, Chernivtsi
  - Teva Investigational Site 5827, Dnipropetrovsk
  - Teva Investigational Site 5828, Donetsk
  - Teva Investigational Site 5829, Ivano-Frankivsk
  - Teva Investigational Site 5830, Kharkiv
  - Teva Investigational Site 5833, Kyiv
  - Teva Investigational Site 5836, Kyiv
  - Teva Investigational Site 5825, Lviv
  - Teva Investigational Site 5839, Odesa
  - Teva Investigational Site 5832, Poltava
  - Teva Investigational Site 5838, Simferopol
  - Teva Investigational Site 5837, Uzhhorod
  - Teva Investigational Site 5826, Vinnytsia
  - Teva Investigational Site 5831, Zaporizhzhya
- United Kingdom (3):
  - Teva Investigational Site 3439, Nottingham
  - Teva Investigational Site 3438, Salford
  - Teva Investigational Site 3440, Sheffield

REFERENCES:
- [Derived] Khan O, Rieckmann P, Boyko A, Selmaj K, Ashtamker N, Davis MD, Kolodny S, Zivadinov R. Efficacy and safety of a three-times-weekly dosing regimen of glatiramer acetate in relapsing-remitting multiple sclerosis patients: 3-year results of the Glatiramer Acetate Low-Frequency Administration open-label extension study. Mult Scler. 2017 May;23(6):818-829. doi: 10.1177/1352458516664033. Epub 2016 Aug 8. PMID 27503905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1524 subjects were screened in this study, and 120 (7.9%) subjects failed screening. Of these, 69 did not meet inclusion or exclusion criteria, 30 withdrew from the study and 21 failed screening for other reasons.
Pre-assignment Details: 1404 subjects were enrolled and randomized in the placebo-controlled (PC) double-blind period. Participants were randomized 2:1 to the treatment arms.
Groups:
- Early Start: GA 40 mg / GA 40 mg: Participants were administered glatiramer acetate (GA) 40 mg/mL by subcutaneous injection three times a week for 12 months during the double-blind Placebo-Controlled Period, and then continued that treatment in the Open-label Period from Month 13 up to Year 6.5 until the study ended.
- Delayed Start: Placebo / GA 40 mg: Participants were administered placebo subcutaneous injections three times a week for 12 months during the double-blind Placebo-Controlled Period. Participants were then switched to glatiramer acetate (GA) 40 mg/mL by subcutaneous injection three times a week during the Open-Label Period from Month 13 up to Year 6.5 until the study ended.
Period: Double-Blind Placebo-Controlled Period
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Started | 943 | 461
Completed | 859 | 430
Not Completed | 84 | 31
Not completed — Death | 0 | 1
Not completed — Adverse Event | 29 | 6
Not completed — Withdrawal by Subject | 34 | 17
Not completed — Physician Decision | 1 | 1
Not completed — Refused to sign informed consent | 4 | 1
Not completed — Noncompliance with study drug | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Pregnancy | 7 | 4
Not completed — Lost to Follow-up | 5 | 1
Period: Open-Label Period
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Started | 834 (Some participants did not continue into the open-label period.) | 419 (Some participants did not continue into the open-label period.)
Completed | 580 | 261
Not Completed | 254 | 158
Not completed — Death | 3 | 1
Not completed — Adverse Event | 30 | 28
Not completed — Withdrawal by Subject | 160 | 88
Not completed — Physician Decision | 13 | 11
Not completed — Non-compliance with study drug | 5 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Pregnancy | 14 | 8
Not completed — Teva requested subject to be withdrawn | 5 | 2
Not completed — Lost to Follow-up | 21 | 20

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) Analysis Set of Participants at the Placebo-Controlled Period Baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg | Total
Number analyzed (Participants) | 943 | 461 | 1404
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.36 (9.401) | 38.12 (9.222) | 37.61 (9.346)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 641 | 313 | 954
  Male | 302 | 148 | 450
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Black or African American | 12 | 3 | 15
  Other, not specified | 12 | 3 | 15
  White | 916 | 455 | 1371
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 934 | 460 | 1394
  Hispanic or Latino | 9 | 1 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant in the Placebo arm was missing the BMI baseline measure.
  kg/m^2
    number analyzed (Participants) | 942 | 461 | 1403
    (all) | 24.38 (4.709) | 24.44 (4.804) | 24.40 (4.739)
Time from First Symptom [Mean (Standard Deviation); unit: years] | 7.68 (6.748) | 7.61 (6.360) | 7.66 (6.621)
Time from Multiple Sclerosis (MS) Diagnosis [Mean (Standard Deviation); unit: years] | 3.70 (4.982) | 3.88 (4.744) | 3.76 (4.904)
Number of T1 Gadolinium (Gd)-Enhanced Lesions per Participant at Baseline [Mean (Standard Deviation); unit: lesions] | 1.7 (4.70) | 1.4 (3.69) | 1.6 (4.39)
Number of T2 Lesions Per Participant at Baseline [Mean (Standard Deviation); unit: lesions] | 38.0 (26.34) | 36.7 (26.68) | 37.5 (26.45)
Sienax Normalized Brain Volume at Baseline [Mean (Standard Deviation); unit: mL] — Sienax estimates total brain tissue volume, from a single image, normalised for skull size. Population: One participant in the GA40 mg ("Early Start') arm was missing the Sienax normalized brain volume baseline measure.
  mL
    number analyzed (Participants) | 942 | 461 | 1403
    (all) | 1533.888 (110.6107) | 1537.899 (110.7549) | 1535.206 (110.6347)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Confirmed Relapses During the Placebo Controlled (PC) Treatment Period Estimated by Negative Binomial Regression
Description: Relapses were monitored throughout the study. During the PC Period, two neurologists/physicians assessed subjects' general medical and neurological evaluations separately. A relapse was defined as the appearance of 1+ new neurological abnormalities or the reappearance of 1+ previously observed neurological abnormalities lasting >= 48 hours and immediately preceded by an improving neurological state of at >=30 days from onset of previous relapse. An event was counted as a relapse only when the subject's symptoms were accompanied by observed objective neurological changes, consistent with >= one of the following: - An increase of >= 0.5 in the Expanded Disability Status Scale (EDSS) score as compared to previous evaluation. - An increase of one grade in the actual score of >=2 of the 7 functional systems (FS), as compared to previous evaluation. - An increase of 2 grades in the actual score of one FS as compared to the previous evaluation. Adjusted mean values are displayed.
Time Frame: Day 1 to 12 months
Population: Intent To Treat (ITT) Analysis Population
Measure: Mean (Standard Error); unit: confirmed relapses
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 943 | 461
confirmed relapses | 0.331 (0.028) | 0.505 (0.049)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Relapses were estimated by a baseline-adjusted, Negative Binomial Regression with an "offset" based on the log of subject's exposure to treatment. The model included the following covariates: - Baseline EDSS score. - Log of the prior 2-year number of relapses. - Volume of T2 lesions at baseliner. - Status of Gd-enhancing T1 activity at baseline (=0 no Gd-enhancing T1 at baseline; =1 at least one Gd-enhancing T1 at baseline). - CGR; Test type: Superiority; p < 0.0001, Negative Binomial Regression — The overall significance level for this study is 5%; Risk Ratio (RR) = 0.656, 95% CI 2-sided [0.539 to 0.799], Standard Error of Mean 0.066 — GA 40 mg vs. placebo

2. Secondary Outcome: The Cumulative Number of New/Enlarging T2 Lesions Taken at Month 6 and Month 12 During the Placebo Controlled (PC) Treatment Period Estimated by Negative Binomial Regression
Description: T2 lesions are hyperintense brain lesions that show on magnetic resonance imaging (MRI) and are associated with multiple sclerosis. The cumulative number of T2 lesions at Months 6 and 12 that are new or enlarged as compared to the baseline MRI are offered. Note that the two timeframes (Months 6 and 12) are combined. Adjusted mean is based on negative binomial regression, adjusted for baseline number of T2 lesions and country or geographical region as covariates.
Time Frame: Baseline (Day -7), Month 6, Month 12
Population: ITT. When a subject had both Month 6 and Month 12 scans missing, the subject was excluded from the analysis. When the Month 12 scan was missing, data from Month 6 was used and an offset of log (0.5) introduced. When the Month 6 scan was missing, data from Month 12 was used with an offset of 0.
Measure: Mean (Standard Error); unit: lesions
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 884 | 441
lesions | 3.650 (0.259) | 5.592 (0.490)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Negative binomial regression; Test type: Superiority; p < .0001, Negative binomial regression — The overall significance level for this study is 5%; Risk Ratio (RR) = 0.653, 95% CI 2-sided [0.546 to 0.780], Standard Error of Mean 0.059 — GA 40 mg vs. placebo

3. Secondary Outcome: The Cumulative Number of Gadolinium (Gd)-Enhanced Lesions on T1-Weighted Images At Month 6 and Month 12 of the Placebo-Controlled (PC) Treatment Period Estimated by Negative Binomial Regression
Description: The cumulative number of gadolinium (Gd)-enhanced lesions on T1-weighted images at Months 6 and 12 as compared to the baseline MRI are offered. Note that the two timeframes (Months 6 and 12) are combined. Adjusted mean is based on negative binomial regression with an "offset" employing the log of the proportion of the number of the available post-baseline scans to adjust for missing MRI scans (if any), adjusted for baseline number of enhancing lesions on T1-weighted images and country or geographical region as covariates.
Time Frame: Baseline (Day -7), Month 6, Month 12
Population: ITT. When a subject had both Month 6 and Month 12 scans missing, the subject was excluded from the analysis.
Measure: Mean (Standard Error); unit: lesions
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 884 | 441
lesions | 0.905 (0.087) | 1.639 (0.194)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Test type: Superiority; p < 0.0001, Negative Binomial Regression — The overall significance level for this study is 5%; Risk Ratio (RR) = 0.552, 95% CI 2-sided [0.436 to 0.699], Standard Error of Mean 0.066 — GA 40 mg vs. placebo

4. Secondary Outcome: Brain Atrophy As Defined by the Percent of Change in Normalized Brain Volume From Baseline to Month 12 During the Placebo Controlled (PC) Treatment Period
Description: The analysis of brain atrophy as defined by the percentage change in normalized brain volume from baseline to Month 12 was based on the outcome of a contrast (GA 40 mg TIW vs. placebo) derived from a baseline-adjusted ANCOVA. In addition to the treatment group, the model included the following covariates: - SIENAX normalized brain volume at baseline. - The number of enhancing lesions on T1-weighted images at baseline. - country or geographical region.
  Sienax estimates total brain tissue volume, from a single image, normalised for skull size.
Time Frame: Baseline (Day -7), Month 12
Population: ITT population of participants who had SIENEX brain volume estimates at both baseline and Month 12.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 840 | 423
percentage change | -0.706 (0.037) | -0.645 (0.047)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Test type: Superiority; p = 0.2058, ANCOVA — The overall significance level for this study is 5%; Mean Difference (Final Values) = -0.061, 95% CI 2-sided [-0.154 to 0.033], Standard Error of Mean 0.048 — GA 40 mg vs Placebo

5. Primary Outcome: Annualized Rate of Confirmed Relapses Comparing Early Starters to Delayed Starters Estimated by Negative Binomial Regression
Description: The annualized relapse rate (ARR) was calculated for the study by dividing the cumulative number of confirmed relapses by the number of person-years of exposure to treatment. The analysis of the annualized relapse rate is based on estimating a contrast (early start vs delayed start) derived from a baseline-adjusted, Negative Binomial Regression model to the number of confirmed relapses observed during study (post randomization) with an "offset" based on the log of exposure to treatment.
Time Frame: Day 1 up to 6.5 years
Population: ITT
Measure: Mean (Standard Error); unit: relapses per year
Groups:
- Early Start: GA 40 mg / GA 40 mg: RParticipants were administered glatiramer acetate (GA) 40 mg/mL by subcutaneous injection three times a week for 12 months during the double-blind Placebo-Controlled Period, and then continued that treatment in the Open-label Period from Month 13 up to Year 6.5 until the study ended.
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 943 | 461
relapses per year | 0.2621 (0.0189) | 0.3146 (0.0279)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Entire Study The Negative Binomial Regression model covariates: • treatment group • PCBL (Placebo-Controlled Baseline) Kurtzke's Expanded Disability Status Scale (EDSS) score as 1 degree of freedom variable • Log of the # of relapses in the 2 years prior to PCBL • Volume of T2 lesions at PCBL • Status of Gd-enhancing T1 lesion activity at PCBL (=0 if no Gd-enhancing T1 lesions at PCBL; =1 if at least one Gd-enhancing T1 lesion at PCBL) • Country or Geographical Region (CGR); Test type: Superiority; p = 0.0409, Negative Binomial Regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.8332, 95% CI 2-sided [0.6995 to 0.9925], Standard Error of Mean 0.0744 — Early Start vs Delayed Start

6. Secondary Outcome: The Number of New/Enlarging T2 Lesions at Months 6, 12 and 36 Estimated by Negative Binomial Regression
Description: All data accumulated from screening, the PC Treatment period up to the end of the Open Label (OL) period are combined and referred to as the Long Term Period. T2 lesions are hyperintense brain lesions that show on magnetic resonance imaging (MRI) and are associated with multiple sclerosis. The number of T2 lesions at Months 6, 12 and 36 that are new or enlarged as compared to the baseline MRI are offered. Adjusted mean is based on negative binomial regression, adjusted for baseline number of T2 lesions and country or geographical region as covariates. An "offset" employing the log of the proportion of the number of the available post-placebo-controlled baseline (PCBL) scans was used to adjust for missing MRI scans.
Time Frame: Baseline (Day -7), Month 6, Month 12, Month 36
Population: ITT population of participants with MRIs at both baseline and the designated timeframes.
Measure: Mean (Standard Error); unit: lesions
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 883 | 440
lesions
  Month 6 | 2.872 (0.214) | 3.902 (0.43)
  Month 12: number analyzed (Participants) | 854 | 425
  Month 12 | 4.484 (0.318) | 7.086 (0.699)
  Month 36: number analyzed (Participants) | 571 | 263
  Month 36 | 5.836 (0.41) | 8.759 (0.82)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 6 Negative binomial regression; Test type: Superiority; p = 0.0056, Negative binomial regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.736, 95% CI 2-sided [0.592 to 0.914], Standard Error of Mean 0.081 — Early Start vs Delayed Start
Statistical Analysis 2: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 12 Negative binomial regression; Test type: Superiority; p < 0.0001, Negative binomial regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.633, 95% CI 2-sided [0.524 to 0.765], Standard Error of Mean 0.061 — Early Start vs Delayed Start
Statistical Analysis 3: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 36 Negative binomial regression; Test type: Superiority; p < 0.0001, Negative binomial regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.666, 95% CI 2-sided [0.557 to 0.797], Standard Error of Mean 0.061 — Early Start vs Delayed Start

7. Secondary Outcome: The Cumulative Number of Gadolinium (Gd)-Enhanced Lesions on T1-Weighted Images At Months 6, 12 and 36 Estimated by Negative Binomial Regression
Description: All data accumulated from screening, the PC Treatment period up to the end of the Open Label (OL) period are combined and referred to as the Long Term Period. The cumulative number of gadolinium (Gd)-enhanced lesions on T1-weighted images at Months 6, 12 and 36 as compared to the baseline MRI are offered. Adjusted mean is based on negative binomial regression The model was fit using an autoregressive covariance structure. Covariates used: number of enhancing lesions on T1-weighted images at placebo-controlled baseline and country or geographical region. The cumulative number is derived from all the data points before it. For example, if the participant skipped one time point in between the baseline and 36 months, then it cannot be calculated.
Time Frame: Baseline (Day -7), Month 6, Month 12, Month 36
Population: ITT population of participants with MRIs at both baseline and the designated timeframes, inclusive of the proceeding post-baseline timeframes.
Measure: Mean (Standard Error); unit: lesions
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 883 | 440
lesions
  Month 6 | 0.629 (0.072) | 1.131 (9.186)
  Month 12: number analyzed (Participants) | 854 | 425
  Month 12 | 1.054 (0.115) | 2.051 (0.282)
  Month 36: number analyzed (Participants) | 570 | 263
  Month 36 | 1.501 (0.168) | 2.265 (0.278)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 6; Test type: Superiority; p = 0.0005, Negative Binomial Regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.556, 95% CI 2-sided [0.4 to 0.773], Standard Error of Mean 0.093 — Early Start vs Delayed Start
Statistical Analysis 2: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 12; Test type: Superiority; p < 0.0001, Negative binomial regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.514, 95% CI 2-sided [0.388 to 0.679], Standard Error of Mean 0.073 — Early Start vs Delayed Start
Statistical Analysis 3: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 36; Test type: Superiority; p = 0.0015, Negative binomial regression — not adjusted for multiplicity; Risk Ratio (RR) = 0.663, 95% CI 2-sided [0.514 to 0.854], Standard Error of Mean 0.086 — Early Start vs Delayed Start

8. Secondary Outcome: Brain Atrophy As Defined by the Percent of Change in Brain Volume From Baseline to Months 6, 12 and 36 Estimated by a Mixed Model for Repeated Measures
Description: The analysis of brain atrophy as defined by the percentage change in brain volume from baseline to Months 6, 12 and 36 was performed using mixed model for repeated measures (MMRM) with SIENAX normalized brain volume at baseline, number of Gd-enhancing lesions at baseline, and country or geographical region as fixed effects.
  Sienax estimates total brain tissue volume, from a single image, normalised for skull size.
Time Frame: Baseline (Day -7), Month 6, Month 12, Month 36
Population: ITT population of participants with SIENEX brain scans at both baseline and the designated timeframes.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: Placebo / GA 40 mg
Number analyzed (Participants) | 872 | 436
percentage change
  Month 6 | -0.429 (0.032) | -0.345 (0.04)
  Month 12: number analyzed (Participants) | 846 | 423
  Month 12 | -0.739 (0.035) | -0.653 (0.046)
  Month 36: number analyzed (Participants) | 543 | 250
  Month 36 | -1.935 (0.063) | -1.952 (0.09)
Statistical Analysis 1: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 6; Test type: Superiority; p = 0.0425, Mixed model for repeated measures (MMRM) — not adjusted for multiplicity; Mean Difference (Final Values) = -0.084, 95% CI 2-sided [-0.166 to -0.003], Standard Error of Mean 0.041 — Early Start vs Delayed Start
Statistical Analysis 2: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 12; Test type: Superiority; p = 0.0844, Mixed model for repeated measures (MMRM) — not adjusted for multiplicity; Mean Difference (Final Values) = -0.086, 95% CI 2-sided [-0.184 to 0.012], Standard Error of Mean 0.05 — Early Start vs Delayed Start
Statistical Analysis 3: Comparison: Early Start: GA 40 mg / GA 40 mg vs Delayed Start: Placebo / GA 40 mg; Month 36; Test type: Superiority; p = 0.8701, Mixed model for repeated measures (MMRM) — not adjusted for multiplicity; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.91 to 0.225], Standard Error of Mean 0.106 — Early Start vs Delayed Start

9. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Early Start: Day 1 up to 6.5 years Delayed Start - Placebo: Day 1 up to Month 12 Delayed Start - GA: Month 13 up to 6.5 years
Population: Glatiramer Acetate (GA) - Treated Analysis Set The GA-Treated analysis set includes all subjects randomized into the study and treated with at least 1 dose of GA at any time during the study. Analyses includes data collected for these subjects from the first time GA was administered.
Measure: Count of Participants; unit: Participants
Groups:
- Delayed Start: GA 40 mg: After completing the double-blind Placebo-Controlled Period, participants had the option of continuing in the study on glatiramer acetate (GA) 40 mg/ml by subcutaneous injection three times a week until the study ended. This 'Delayed Start' treatment began at Month 13 and continued until the study ended (up to about 6.5 years).
- Delayed Start: Placebo: Participants were administered placebo subcutaneous injections three times a week from Day 1 to Month 12 during the double-blind Placebo-Controlled Period.
Arm/Group | Early Start: GA 40 mg / GA 40 mg | Delayed Start: GA 40 mg | Delayed Start: Placebo
Number analyzed (Participants) | 943 | 419 | 461
Participants
  Any TEAE | 777 | 322 | 284
  Severity of TEAEs: Mild | 698 | 283 | 247
  Severity of TEAEs: Moderate | 441 | 168 | 101
  Severity of TEAEs: Severe | 95 | 24 | 16
  Treatment-related TEAEs | 501 | 189 | 73
  Serious TEAEs | 117 | 36 | 21
  Deaths | 3 | 1 | 1
  TEAEs leading to treatment discontinuation | 63 | 28 | 6

ADVERSE EVENTS:
Time Frame: Delayed Start (GA 40 mg): Month 13 up to 6.5 years Delayed Start (Placebo): Day 1 to Month 12 Early Start: (GA 40 mg/ GA 40 mg) Day 1 up to 6.5 years
Description: Death details:
  Delayed Start (GA 40 mg): caused by subarachnoid hemorrhage and brain edema 1027 days after the first dose of GA.
  Delayed Start (Placebo): cardiopulmonary failure
  Early Start: Three deaths due to acute cardiac failure, cardio-respiratory arrest, and cardiac arrest occurring 488, 1283 and 1682 days after first dose of GA respectively.
Groups:
- Delayed Start: GA 40 mg: After completing the double-blind Placebo-Controlled Period, participants had the option of continuing in the study on glatiramer acetate (GA) 40 mg/ml by subcutaneous injection three times a week until the study ended. This 'Delayed Start' treatment started at Month 13 and continued until the study ended (up to about 6.5 years).
Arm/Group | Delayed Start: GA 40 mg | Delayed Start: Placebo | Early Start: GA 40 mg / GA 40 mg
All-Cause Mortality (participants affected / at risk) | 1/419 | 1/461 | 3/943
Serious Adverse Events (participants affected / at risk) | 36/419 | 21/461 | 117/943
Other Adverse Events (participants affected / at risk) | 238/419 | 167/461 | 609/943
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Start: GA 40 mg (N=419) | Delayed Start: Placebo (N=461) | Early Start: GA 40 mg / GA 40 mg (N=943)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 2 (4)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (3)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Immediate post-injection reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (3) | 0 (0) | 1 (2)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Burn infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gallbladder empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured skull depressed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 4 (4)
Apallic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Multiple sclerosis relapse (Nervous system disorders) | 2 (3) | 1 (1) | 5 (5)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Perinephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine cervical erosion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Breast conserving surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cervix operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 2 (3) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Ureteric calculus removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Start: GA 40 mg (N=419) | Delayed Start: Placebo (N=461) | Early Start: GA 40 mg / GA 40 mg (N=943)
Injection site erythema (General disorders) | 107 (122) | 8 (10) | 243 (391)
Injection site pain (General disorders) | 55 (61) | 10 (10) | 115 (138)
Injection site pruritus (General disorders) | 23 (24) | 2 (2) | 68 (95)
Injection site swelling (General disorders) | 23 (23) | 3 (5) | 50 (95)
Bronchitis (Infections and infestations) | 20 (25) | 7 (9) | 50 (65)
Influenza (Infections and infestations) | 25 (33) | 17 (22) | 67 (103)
Nasopharyngitis (Infections and infestations) | 56 (98) | 39 (47) | 167 (346)
Upper respiratory tract infection (Infections and infestations) | 32 (54) | 25 (30) | 98 (158)
Urinary tract infection (Infections and infestations) | 36 (50) | 22 (24) | 103 (165)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (45) | 20 (26) | 98 (150)
Headache (Nervous system disorders) | 39 (83) | 55 (71) | 132 (316)
Multiple sclerosis relapse (Nervous system disorders) | 10 (12) | 7 (9) | 48 (63)

LIMITATIONS AND CAVEATS:
Analyses of Open-Label Period data are not adjusted for multiplicity and therefore do not control for type one statistical error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.